CLINICAL TRIAL: NCT01973075
Title: Genetic Etiology in Premature Ovarian Insufficiency
Acronym: POI
Status: Completed | Type: Observational
Sponsor: BEGUM AYDOGAN (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Sponsor-Investigator, BEGUM AYDOGAN, MD,OBGYN, Sisli Hamidiye Etfal Training and Research Hospital
Organization: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Other Study IDs: 22547
Record Dates: First submitted 2013-10-20; First posted 2013-10-31 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Primary Ovarian Insufficiency; Genetic Predisposition to Disease
Keywords: Premature Ovarian Insufficiency (POI)
MeSH Terms: conditions — Primary Ovarian Insufficiency; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — 4ml whole blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- premature ovarian Insufficiency: 4ml whole blood sample is going to collect from premature ovarian Insufficiency group for the assessment of genetic abnormalities
- healthy control group: 4 ml of whole blood is going to taken from healthy control group

SUMMARY:
Premature Ovarian Insufficiency (POI), first described by Albright in 1942, is defined as an increase in Follicle Stimulating Hormone (FSH), an insufficiency of the ovarian function leading to an early menopause (<40 years of age).Today, only 35% of POI's etiology can be explained. Causes enlightening POI may be enumerated as follows, according to their frequency: genetic mutations, autoimmune defects and abnormalities detected on the X chromosome.The purpose of the study is to determine the frequency of the genetic abnormalities and polymorphisms described above in the POI Turkish population

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosed premature ovarian failure patients
* 20-40 years old female patients

Exclusion Criteria:

* Surgical surgical menopause
* Female patients who can't meet the age range criteria

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients who are admitted to obstetrics and gynecology department
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2016-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Genetic etiology in Premature ovarian Insufficiency | up to 1 year
  In the framework of our project, abnormalities on the X chromosome will be studied by karyotyping, follicle-stimulating hormone receptor (FSHR),nuclear receptor subfamily 5,group A,member 1 (NR5A1),Newborn ovary homeobox gene (NOBOX),Bone morphogenetic protein 15 (BMP15) genes will be analyzed by sequencing and finally repeat size analysis for FMR1 gene will be performed fragment analyses, on 75 POI and 25 healthy control population.Collected data will enable us to determine the frequency of the abnormalities and polymorphisms described above in the POI Turkish population. Patients free of those genetic variants will help us to identify new loci or genes implicated in POI.

CONTACTS AND LOCATIONS:
Overall Officials: Engin Oral, Prof,OBGYN, Study Director — Istanbul University
Locations (1):
- Istanbul University Cerrahpasa Medical school Obstetrics department, Istanbul, Turkey (Türkiye)